CLINICAL TRIAL: NCT05763563
Title: Feasibility Of Exercise Prehabilitation Among Older Patients With Hematological Malignancies Preparing For Chimeric Antigen Receptor (CAR) T-Cell Immunotherapy
Brief Title: Exercise Prehabilitation Among Older Patients With Hematological Malignancies Preparing For CAR-T Cell Immunotherapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Cancer and Aging Research Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-22115
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma; Leukemia; Myeloma
MeSH Terms: conditions — Lymphoma; Leukemia; Neoplasms, Plasma Cell | interventions — Resistance Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise prehabilitation (Experimental): Participants will take part in an exercise program in which they will be encouraged to perform approximately 30 minutes of resistance training exercises approximately twice per week until they undergo CAR-T therapy (Approximately 4-6 weeks). Participants will also be encouraged to perform moderate aerobic exercise such as brisk walking or using stationary aerobic equipment at least 3 times per week. Participants will wear a FitBit fitness watch to monitor aerobic exercise.
  Interventions: Behavioral: Resistance Training; Behavioral: Aerobic Exercise; Behavioral: Optional Aerobic Exercise Procedure; Radiation: Optional In-Person Exercise Sessions

INTERVENTIONS:
Behavioral: Resistance Training — Participants will be encouraged to perform approximately 30 minutes of resistance training exercises twice per week, until they undergo CART-T therapy. Exercises will be performed using resistance tubes (Bodylastics Resistance Bands Set) and a connectable bar (Bionic Body Workout Bar) that mimics a weighted barbell when tubes are attached. The tubes provide up to 142 pounds of resistance (adjustable in increments between 3-10 pounds) when simultaneously connected to handles or bar, and multiple tubes can be attached simultaneously.
Behavioral: Aerobic Exercise — Participants will be encouraged to perform ≥30 minutes of moderate-intensity aerobic exercise on ≥3 days per week. Aerobic exercise intensity will be guided by heart rate zones, with participants exercising at 50-70% of their age-predicted maximum heart rate in bouts of at least 10 minutes at a time. Participants will be encouraged to gradually increase exercise intensity and duration until they are meeting the recommendation
Behavioral: Optional Aerobic Exercise Procedure — Participants will be encouraged to complete 3 tele-supervised aerobic training sessions per week, each lasting 30 minutes. Participants will be encouraged to achieve moderate exercise intensity based on heart rate visualized on PM5 monitors. Participants will report their heart rates every 3-5 minutes during an exercise session and be encouraged to adjust pedaling cadence or flywheel resistance accordingly to achieve moderate intensity.
  Exercise trainers will access logged heart rate ranges (64-76% of age-predicted maximum heart rate) to provide individualized and appropriate guidance during sessions.
  Participants who are untrained or otherwise uncomfortable maintaining moderate aerobic intensity for 30 minutes will be encouraged to gradually increase the duration and intensity of their sessions until they are meeting these guidelines.
Radiation: Optional In-Person Exercise Sessions — Participants who prefer to complete RT and/or aerobic exercise sessions in-person will be allowed to do so. These sessions will be conducted in the Moffitt Promotes Resilience in Oncology Via Exercise (MPROVE) Laboratory using the same equipment participants would use for Zoom sessions, with guidance and supervision from certified exercise trainers.

SUMMARY:
The purpose of the study is to evaluate an exercise program for individuals preparing for Chimeric Antigen Receptor (CAR) T-cell immunotherapy for hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Lymphoma, leukemia, or myeloma with commercial FDA-approved CAR-T delivery planned for ≥4 weeks following enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Able to read and speak English fluently
* Capable of providing informed consent
* For optional, tele-supervised aerobic training procedure involving stationary bicycle delivery, participants must live within a 2-hour drive of Moffitt Cancer Center as determined via Google Maps.

Exclusion Criteria:

* Regular engagement in Resistance training (2x/week targeting all major muscle groups)
* Screen failure for exercise safety based on Physical Activity Readiness Questionnaire (PAR-Q) and Patient-Reported Measurement Information System (PROMIS) screening questions
* Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease (New York Heart Association functional class III or IV).
* Recent fracture or acute musculoskeletal injury that precludes ability to participate in RT using body weight
* Numeric pain rating scale of ≥ 7 out of 10
* Myopathic or rheumatologic disease that impacts physical function
* Cognitive, visual, or auditory limitations that preclude safe engagement in remotely-supervised resistance training sessions or independent aerobic exercise (as determined by patients' treating oncologists and specified in clinic notes outlining disease history).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants that Enroll and Consent - Enrollment Feasibility | Up to 12 Months
  Enrollment will be considered feasible if ≥60% of eligible and approached patients actually consent and enroll
Percentage of Participants that Complete Study Assessments - Retention Feasibility | Up to 3 Months
  Retention will be considered feasible if ≥70% of participants complete study measures
Adherence - Feasibility | Up to 3 Months
  Adherence will be based on participants attending ≥ 70% of tele-RT sessions on average and performing ≥ 70% of prescribed moderate-intensity aerobic exercise per week
Participant Evaluation of Feasibility and Acceptability - Acceptability | Up to 3 Months
  Participants evaluation of feasibility and acceptability will be assessed with a questionnaire, adapted to fit the intervention. The questionnaire includes both Likert Scale and open-ended questions. An item-by-item basis and as average item score, with scores ≥4 ("agree" to "strongly agree") indicating acceptability. Open-ended responses will be analyzed qualitatively to inform intervention improvement.
Participant Self-Reported Musculoskeletal Injuries - Safety | Up to 3 Months
  The numerator of the safety variable will be the number of musculoskeletal injuries or adverse health events reported as "likely related" or "definitely related" the exercise programming and that caused at least some limitation of daily activity lasting more than 3 days. The denominator of the safety variable will be the number of exercise sessions performed by the participant (tele-resistance training plus aerobic exercise sessions lasting ≥10 minutes). The intervention will be considered safe if the rate of musculoskeletal injuries (i.e., muscle strains or pulls, sprains, exacerbated bone pain, fractures or breaks, or other adverse health events incurred during exercise sessions) is lower than the published metric of 11.9 injuries per 1000 sessions, as used as a benchmark in previous exercise oncology research
Objective physical functioning and fitness - Baseline | At Baseline
  Physical functioning and fitness will be assessed using the 30-second chair stand test,30-second arm curl test, and treadmill 6-minute walk test.
Objective physical functioning and fitness - Follow-up | Up to 3 Months
  Physical functioning and fitness will be assessed using the 30-second chair stand test,30-second arm curl test, and treadmill 6-minute walk test.
Participant Skeletal Muscle Index (SMI) - Baseline | Baseline
  Participants SMI will be measured using Tomovision SliceOMatic software and clinical, computerized tomography (CT) scans
Participant Skeletal Muscle Index (SMI) - Follow-up | After CAR-T Therapy, Up to 6 Months
  Participants SMI will be measured using Tomovision SliceOMatic software and clinical, computerized tomography (CT) scans
Participants Health-Related Quality of Life - Baseline | Baseline
  Participants health-related quality of life will be measured using the 12-item Medical Outcomes Study Short Form Survey
Participants Health-Related Quality of Life - At 3 Months | Up to 3 Months
  Participants health-related quality of life will be measured using the 12-item Medical Outcomes Study Short Form Survey
Participants Health-Related Quality of Life - At 6 Months | Up to 6 Months
  Participants health-related quality of life will be measured using the 12-item Medical Outcomes Study Short Form Survey
Participant Self Reported Exercise - Baseline | Baseline
  Participant self-reported exercise will be measured using a modified Godin Leisure Time Exercise Questionnaire to assess both aerobic and resistance exercise
Participant Self Reported Exercise - At 3 Months | Up to 3 Months
  Participant self-reported exercise will be measured using a modified Godin Leisure Time Exercise Questionnaire to assess both aerobic and resistance exercise
Participant Self Reported Exercise - At 6 Months | Up to 6 Months
  Participant self-reported exercise will be measured using a modified Godin Leisure Time Exercise Questionnaire to assess both aerobic and resistance exercise

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Parker, PhD, MPH, Principal Investigator — Moffitt Cancer Center; Ciara Freeman, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinicaltrialssearch?DiseaseSite=&q=22115